CLINICAL TRIAL: NCT06361199
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Phase Ib Study to Evaluate the Tolerability, Pharmacokinetics and Pharmacodynamics of Proximod in Healthy Subjects and Patients With Rheumatoid Arthritis.
Brief Title: Proximod Pharmacokinetics in Healthy Subjects and Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longevity Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJXH-2021-001
Record Dates: First submitted 2024-03-12; First posted 2024-04-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, qd, oral administration for 28 days
  Interventions: Drug: Placebo
- Proximod (Experimental): Proximod Tablets, 5mg, qd, oral administration for 28 days
  Interventions: Drug: Proximod

INTERVENTIONS:
Drug: Proximod — Multiple-dose to establish the safety and PK profile in both healthy subjects and patients with rheumatoid arthritis
  Other Names: IMM-H001
  Arms: Proximod
Drug: Placebo — Placebo controlled
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the tolerability, pharmacokinetics and pharmacodynamics of Proximod in healthy subjects and patients with rheumatoid arthritis. The main questions it arms to answer are:

1. to evaluate the safety and tolerance of Proximod in health subjects after repeated doses.
2. to assess the pharmacokinetics and pharmacodynamics of Proximod in healthy subjects after repeated doses.
3. to evaluate the safety and tolerance of Proximod in patients with rheumatoid arthritis.
4. to evaluate the pharmacokinetics and pharmacodynamics of Proximod in patients with rheumatoid arthritis.

Participants will receive test tablets or placebo at the indicated date and collect blood samples.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Before the test, sign an informed consent form and fully understand the written test content, process and possible adverse reactions.
* Complete research in accordance with the requirements of the trial plan.
* Subjects (including partners) are willing to have no pregnancy plans in the next 6 months and voluntarily take effective contraceptive measures.
* Male and female subjects aged 18 to 50 years old (including 18 and 50 years old).
* Male subjects must weigh no less than 50 kg, and female subjects must weigh no less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), body mass index is in the range of 18~28kg/m2 (including the critical value).
* Health status: No clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system (such as asthma, exercise-induced asthma, chronic obstructive pulmonary disease), mental disorder, metabolic abnormality, etc.
* Normal physical examination and vital signs or abnormal without clinical significance.

Exclusion Criteria for healthy subjects:

* Those who smoked more than 5 cigarettes per day in the 3 months before the test.
* Have a history of allergy to the trial drug or its excipients, or allergic constitution (allergy to multiple drugs and food).
* Have a history of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine).
* Blood donation or significant blood loss (>450 mL) within three months before screening.
* Taking any drugs that alter liver enzyme activity 28 days before screening.
* Take any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines within 14 days before screening.
* Those who have taken special diets (including dragon fruit, mango, grapefruit, etc.) or engaged in strenuous exercise within 2 weeks before screening, or other factors that affect drug absorption, distribution, metabolism, excretion, etc.
* Recent significant changes in eating or exercise habits.
* Participated in a drug clinical trial within three months before taking the study drug.
* Have a history of dysphagia or any gastrointestinal disease that affects drug absorption.
* Suffering from any disease that increases the risk of bleeding, such as acute gastritis or gastric and duodenal ulcers.
* ECG abnormalities have clinical significance or QTC>470ms in men or QTC>480ms in women.
* Abnormal ophthalmic examination with clinical significance, including fundus examination and optical coherence tomography.
* Those who have a history of uveitis and are not suitable to participate in the trial as considered by the researcher.
* Those who have a history of herpes zoster or chickenpox.
* Female subjects are lactating or have positive serum pregnancy results during the screening period or during the trial.
* Clinically significant abnormalities in clinical laboratory tests or other clinically significant following diseases diagnosed within 12 months (including but not limited to gastrointestinal, renal, liver, neurological, blood, endocrine, tumor, lung, immune, psychiatric or Cardiovascular disease).
* Positive screening results for viral hepatitis (including hepatitis B and hepatitis C), HIV antibodies, and Treponema pallidum antibodies.
* Acute illness or concomitant medication occurs from the screening stage to study medication.
* Ingested chocolate, any caffeinated or xanthine-rich food or drink 24 hours before taking study drug.
* Positive alcohol breath test 24 hours before taking study medication or upon - Those with a positive urine drug screen or those with a history of drug abuse in the past five years or those who have used drugs 3 months before the test.
* Subjects who the researcher believes have other factors that are not suitable for participating in this trial.

Inclusion Criteria for patients with rheumatoid arthritis:

* Sign an informed consent form before the trial and fully understand the trial content, process and possible adverse reactions.
* Age ranges from 18 to 70 years old (both ends included), regardless of gender;
* Male subjects must weigh no less than 50 kg, and female subjects must weigh no less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), body mass index is in the range of 18~30 kg/m2 (including the critical value).
* Subjects (including partners) are willing to voluntarily take effective contraceptive measures within 6 months from screening to the last dose of study drug.
* Diagnosed with rheumatoid arthritis, using the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria .
* C-reactive protein or high-sensitivity C-reactive protein (CRP/hsCRP) ≥ the upper limit of normal value during screening.
* Have not used any disease-modifying antirheumatic drugs (DMARDs) before the first dose of the trial, or have used methotrexate (MTX) at a stable dose for ≥4 weeks before the first dose, or have used methotrexate, Those who have stopped taking sulfasalazine, chloroquine/hydroxychloroquine, gold preparations, penicillamine and other drugs for ≥7 drug half-lives before the first dose.
* The subjects can communicate well with the researchers, understand and comply with the requirements of this study, and can complete the experiment in accordance with the requirements of the trial protocol.

Exclusion Criteria for patients with rheumatoid arthritis:

* Those who are allergic to the main ingredients and excipients of Prosemod tablets, or have allergies (allergic to multiple drugs and food).
* Have any diseases that may affect the absorption of the drug in the body, such as dysphagia or gastrointestinal system diseases.
* Abnormal eye examinations with clinical significance, including fundus examination and optical coherence tomography.
* Any laboratory test indicator during screening or baseline examination meets the following standards:

AST or ALT>1.5 times ULN Total bilirubin>2 times ULN Hemoglobin (male) <10.0g/dL (100.0g/L), or (female) <9.0g/dL (90.0g/L) Total white blood cell count <3.0×109/L Neutrophil count <1.0×109/L Creatinine clearance rate (CLcr) ≤50 mL/min Any clinically significant laboratory abnormal values that the researcher believes may interfere with the evaluation of the results of this study.

* QTC during the electrocardiogram during the screening period is > 470 ms for men and > 480 ms for women, or those who are judged by the researcher to be abnormal and clinically significant and who judge that they cannot be enrolled.
* Those who screen positive for viral hepatitis (including hepatitis B and hepatitis C), HIV antibodies, and Treponema pallidum antibodies (positive Treponema pallidum patients need to be tested for RPR, and the researcher will decide whether to be included based on the results), or those who are negative for hepatitis B surface antigen and have hepatitis B surface antigen Antibody negative, hepatitis B core antibody positive and HBV DNA quantification >0.
* Female subjects who are lactating or have positive serum pregnancy results during the screening period or trial, or who plan to become pregnant or breast-feeding during the study or within 6 months after the last dose.
* Those with positive urine drug screening and alcohol breath tests.
* Have a history or evidence of any of the following diseases:

Those with any systemic inflammatory disease except RA. People with Felty syndrome. Decompensated heart failure (New York Heart Association classification III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistent and Clinically significant arrhythmias, coronary artery bypass grafting, or percutaneous coronary intervention.

Have a history of lymphoproliferative disease, or have various signs or symptoms that may be lymphoproliferative disease, including lymphadenopathy or splenomegaly, or have experienced treated or untreated malignant tumors, whether localized or not Evidence of recurrence or metastasis.

The subject has any active malignant tumor or history of malignant tumor within 5 years before the screening visit, except for cutaneous squamous or basal cell carcinoma, cervical carcinoma in situ, or breast ductal carcinoma in situ that has been treated and considered cured .

Suffer from genetic immunodeficiency or have a family history of hereditary immunodeficiency.

Those who have a history of uveitis and are not suitable to participate in the trial as considered by the researcher.

Those who have undergone joint surgery within 6 months before the first dose of the trial.

Those who have severe infection within 3 months before screening or acute infection symptoms within 7 days before screening are judged by the researcher to be unsuitable participants.

Those who have a history of herpes zoster or chickenpox. Those who have a history of drug abuse or have used drugs within the past five years.

Have cardiovascular, respiratory system, liver, kidney, digestive tract, immune, blood, endocrine, metabolic, psychiatric and neurological diseases or history, which may affect the absorption, distribution, metabolism and excretion of the drug or interfere with the results according to the researcher's judgment evaluator.

10. Use of any of the following drugs or treatments: Received intra-articular, intramuscular injection, intravenous injection, trigger point or tender point, intracapsular, or intratendinous glucocorticoid treatment within 8 weeks before the first dose.

Those who have used any non-steroidal anti-inflammatory drugs (NSAIDs) or oral corticosteroids within 1 week before the first dose of the trial.

Received iguratimod or interferon treatment (such as Lusperin, Ganlenon, Rebetron, etc.) within 1 month before the first dose.

Those who have received any live vaccine, attenuated vaccine or inactivated vaccine within 1 month before the first dose (for example, those who have received the new coronavirus vaccine need to wait 4 weeks or more after completing the last dose before they can be enrolled).

Have used other drugs known to have strong immunosuppressive or immunomodulatory effects (such as Pavlin, Tripterygium wilfordii, Mycophenolate mofetil, Cyclospora) within 4 weeks before the first dose. (e.g., tacrolimus, azathioprine, 6-mercaptopurine, etc.).

Those who have used any other prescription drugs, over-the-counter drugs, Chinese herbal medicines, food or food supplements that may have an impact on the test drug, such as CYP3A4 inhibitors or inducers, within 2 weeks before the first dose of the trial. , grapefruit juice, etc.

* Those who smoke, drink alcohol, or drink food and beverages containing xanthine or caffeine, exercise strenuously, or have other factors that affect drug absorption, distribution, metabolism, excretion, etc. 2 days before the first dose of the test.
* Those who have participated in any clinical trials of drugs or medical devices within 1 month before screening.
* Those who donated blood or suffered massive blood loss (>450 mL) within three months before screening, or those who intend to donate blood during the study or within 1 month after the end of the study.
* Subjects who the researcher believes have other factors that are not suitable for participating in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 48 days
Time to peak plasma concentration (Tmax) | Up to 48 days
The lowest plasma concentration (Cmin) | Up to 48 days
Half-life (t1/2) | Up to 48 days
Area under the plasma concentration versus time curve (AUC) | Up to 48 days
Number of adverse events and number of participants with adverse events | Up to 48 days

SECONDARY OUTCOMES:
Lymphocyte count | Up to 48 days
Percentage of CD3+CD4+ and CD3+CD8+T cells | Up to 48 days
ACR20 score in Patients With Rheumatoid Arthritis | Day 8, 15, 22, 29 and 48 compared to baseline
Disease Activity Score（DAS28-CRP）in Patients With Rheumatoid Arthritis | Day 8, 15, 22, 29 and 48 compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Li Q, Li C, Wu M, Chen H, Li Y, You F, Zhao Y, Jin J, Chen X, Ding Y. Evaluation of proximod, a selective agonist of sphingosine-1-phosphate receptor-1, in healthy volunteers and patients with rheumatoid arthritis: a phase 1, double-blind, randomised, placebo-controlled, ascending dose trial. Lancet Rheumatol. 2024 Dec;6(12):e837-e847. doi: 10.1016/S2665-9913(24)00199-1. Epub 2024 Oct 22. PMID 39454617